CLINICAL TRIAL: NCT05117567
Title: A Personal Protection Package for Reducing Malaria Transmission in Forest-going Mobile and Migrant Populations in Lao PDR and Cambodia: A Stepped-wedge Trial With Nested Mixed-methods Study
Brief Title: Reducing Malaria Transmission in Forest-going Mobile and Migrant Populations in Lao PDR and Cambodia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Health Poverty Action (Other); Centre of Malariology Parasitology and Entomology, Department of Communicable Diseases Control, Ministry of Health, Lao PDR (Unknown); National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 388/21_forest_Cambodia_Laos
Record Dates: First submitted 2021-08-16; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Plasmodium Infection
Keywords: malaria; prevention; vector; migrant; elimination; vivax; falciparum; community-delivered; intervention
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized controlled trial (one-way crossover) with nested mixed methods study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal protection package (Experimental): A personal protection package that includes Long-lasting insecticidal hammock net (LLIHN), insect repellent (Icaridin), and mobile and migrant population-tailored behavioural change communication (BCC) package
  Interventions: Combination Product: Personal protection package
- Control (No Intervention): No personal protection package

INTERVENTIONS:
Combination Product: Personal protection package — A personal protection package that includes Long-lasting insecticidal hammock net (LLIHN), insect repellent (Icaridin), and MMP-tailored behavioural change communication (BCC) package
  Arms: Personal protection package

SUMMARY:
This stepped-wedge cluster-randomized controlled trial with nested mixed methods study will assess the effectiveness, acceptability, feasibility and cost-effectiveness of a personal protection package to reduce malaria transmission among mobile and migrant populations (MMPs) and the general population in their residing villages in Lao People's Democratic Republic (PDR) and Cambodia.

DETAILED DESCRIPTION:
Over the last decade, the burden of malaria has fallen dramatically in the Greater Mekong Subregion, with deaths falling by 95% and cases by 76% between 2012 and 2019.The declining malaria burden in GMS has largely attributed by the deployment of interventions of malaria prevention tools such as long-lasting Insecticidal Nets (LLIN), and widespread availability of rapid diagnostic tests and artemisinin combination therapies. However, residual transmission still exists among high risk populations, particularly mobile and migrant populations who enter forests for work. New interventions targetting these high risk groups are needed if countries of the Greater Mekong Subregion are to achieve malaria elimination by 2030. The study will be conducted in malaria endemic areas of Lao PDR (Attapeu, Saravanh, Savannakhet and Khammouane Provinces) and Cambodia (Preah Vihear, Stung Treng and Ratanakiri Provinces) which have large forest going MMP populations. The aim of the study is to assess the effectiveness, acceptability, feasibility and cost-effectiveness of a personal protection package to reduce malaria transmission among mobile and migrant populations (MMPs) and the general population in their residing villages in Lao People's Democratic Republic (PDR) and Cambodia. The personal protection package comprises a long-lasting insecticidal hammock net (LLIHN), insect repellent (Icaridin), and a behavioural change communication (BCC) package tailored to mobile and migrant populations. The study design is a stepped-wedge cluster-randomized controlled trial with nested mixed methods study. The stepped-wedge cluster randomized trial will estimate the effectiveness of a personal protection package provided to forest-going MMPs (the intervention) delivered by village malaria volunteers at the site (village/worksite) level on reducing Plasmodium spp. infections. Whilst the personal protection package will be provided to mobile and migrant populations in each village in a step-wise manner, primary and secondary outcomes relating to malaria testing will be collected in all consenting individuals in the village who present for malaria rapid diagnostic tests, whether they are mobile and migrant people or not.

The open stepped-wedge cluster-randomised controlled trial, randomized at the volunteer level (i.e. the volunteer and the village / workplaces they service), will be implemented between July 2021 to June 2022. The personal protection package for MMPs will be implemented sequentially in a minimum of ~488 villages serviced by approximately ~488 VMWs (~428 in Lao PDR and ~60 in Cambodia). Villages from each country will be randomised into 11 ordered blocks, with blocks transitioned from control (no personal protection package) to intervention (distribution of personal protection package) states at monthly intervals (10 blocks of 44 villages for the first 10 steps and a block of 48 villages transitioned at the last step). This follows an initial baseline control period of one-month at the start of the study

Approximately 11 RDTs per month will be undertaken in each study site (village/ worksite). Given the design we estimate that the study has power to detect a relative minimum detectable difference of 34% (OR = 0.66) in odds of RDT-detectable malaria infection due to the intervention (assuming a village intraclass correlation [ICC]= 0.42; 5% significance; 90% power and 1% RDT malaria prevalence).

For the stepped-wedged cluster randomized trial, both descriptive and primary outcome trial analyses will be performed. Using Stata version 15, differences in prevalence of Plasmodium spp. infections will be estimated across intervention and control periods using generalized linear mixed modelling (e.g. logit link function and binomial distribution) with crossed random effects for village and time, and intervention state, time and seasonality estimated as independent fixed factors. Temporal and spatial trends of Plasmodium spp. infections will also be explored including analysis of the effectiveness of the intervention across the study period. We will also explore any village-specific heterogeneity in effect by specifying a random effect for the intervention. Generalised linear mixed modelling will be extended to include model terms for country (main and interaction effects), and these will used to assess the extent of country-specific heterogeneity in intervention effect. The same approach will be used to assess risk group-specific heterogeneity (MMP, forest-goer, villager) in intervention effect.

ELIGIBILITY:
Inclusion:

Mobile and migrant individuals aged 18 years and over in selected villages including:

* Traditional slash-and-burn and paddy field farming communities visiting their forest farms (commonly ethnic minority groups)
* Seasonal agricultural laborers
* Forest workers in the informal sector (hunters, small-scale gem/gold miners, people gathering forest products (precious timber, construction timber, rattan/bamboo)
* Transient or mobile camp residents associated with commercial projects (road/pipeline construction, large-scale logging, deep seaport projects, etc.)
* Formal and informal cross-border migrant workers

For qualitative research component, local health stakeholders meeting the following criteria will be eligible:

* Aged 18 years and over
* The local health stakeholders such as health centre staff, Operational District Malaria Supervisor (ODMS), and Provincial Malaria Supervisor (PMS), and basic health staff such as malaria unit staff in health centres, midwives, health assistants, district health officers and district focal person from CMPE and CNM
* Health staff members from HPA and Lao malaria community service organisations

Exclusion:

A village will be excluded from the study if:

The village has an VHV/VMW program operated by any organizations other than CMPE, CNM, HPA, malaria CSOs in Lao PDR The village has no malaria cases or API less than 1 in any of the past three years (2018 - 2020) The village has no MMPs The village has no VHV/VMW The village has a government health facility for provision of malaria services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5868 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Plasmodium spp. infection diagnosed by RDT | Assessed weekly, longitudinally over 12 months
  Change in the number of Plasmodium spp. infections detected by RDT per week per village

SECONDARY OUTCOMES:
Symptomatic malaria diagnosed by RDT | Assessed weekly, longitudinally over 12 months
  Change in the number of symptomatic Plasmodium spp. infections detected by RDT per week per village
Plasmodium spp. infection as determined by polymerase chain reaction (PCR) on RDT cassette samples | Assessed weekly, longitudinally over 12 months
  Change in the prevalence of Plasmodium spp. infection as determined by polymerase chain reaction (PCR) from RDT cassette samples
Plasmodium spp. infection as determined by polymerase chain reaction (PCR) on dried blood spot samples | Assessed weekly, longitudinally over 12 months
  Change in the prevalence of Plasmodium spp. infection as determined by polymerase chain reaction (PCR) from dried blood spot (DBS) samples
Plasmodium spp. infections with drug resistance mutations | Assessed weekly, longitudinally over 12 months
  Change in the prevalence of Plasmodium spp. infection with drug resistance mutations.
Prevalence of antibodies to Plasmodium spp. | Assessed weekly, longitudinally over 12 months
  Prevalence of antibodies to Plasmodium spp. determined by Enzyme Linked Immunosorbent assay (ELISA) from RDT and DBS samples
Levels of antibodies to Plasmodium spp. | Assessed weekly, longitudinally over 12 months
  Levels of antibodies to Plasmodium spp. determined by Enzyme Linked Immunosorbent assay (ELISA) from RDT and DBS samples
Prevalence of antibodies to vector salivary antigens | Assessed weekly, longitudinally over 12 months
  Levels of antibody biomarkers of vector exposure
Levels of antibodies to vector salivary antigens | Assessed weekly, longitudinally over 12 months
  Levels of antibody biomarkers of vector exposure
Levels of knowledge, attitude and practice regarding malaria prevention among MMPs | At approximately 12 months
  Focus group discussions
Proportion of survey respondents (MMPs) who accept and are willing to use/ did use the personal protection package according to the protocol | At approximately 12 months
  Questionnaire

REFERENCES:
- [Derived] Gabaldon Figueira JC, Wagah MG, Adipo LB, Wanjiku C, Maia MF. Topical repellents for malaria prevention. Cochrane Database Syst Rev. 2023 Aug 21;8(8):CD015422. doi: 10.1002/14651858.CD015422.pub2. PMID 37602418
- [Derived] Htike W, Oo WH, Lynn T, Sovanda L, Agius PA, Oo MC, Galau NH, Thu KM, Zaw AK, Htwe EP, Cutts JC, Kearney EA, Scott N, O'Flaherty K, Wang B, Khamlome B, Vilay P, Siv S, Fowkes FJI. Reducing malaria transmission in forest-going mobile and migrant populations in Lao PDR and Cambodia: protocol for stepped-wedge cluster-randomised controlled trial. BMC Infect Dis. 2022 Sep 24;22(1):747. doi: 10.1186/s12879-022-07724-5. PMID 36153501